CLINICAL TRIAL: NCT01771276
Title: Evaluating Impact of ULTIMATE Number of G-CATH EZ- Suture Anchors Placed Endoscopically on Motility, Metabolism, Satiety, and Weight Utilizing the Incisionless Operating Platform for the Treatment of Primary Obesity
Brief Title: ULTIMATE Study for Weight Loss
Acronym: ULTIMATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USGI Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPR602
Record Dates: First submitted 2012-09-04; First posted 2013-01-18 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: POSE
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultimate Anchor (Experimental): Use of the g-Cath Suture Anchor Delivery Catheter and accessories in placing the ultimate number of anchors for weight loss.
  Interventions: Device: g-Cath Suture Anchor Delivery Catheter

INTERVENTIONS:
Device: g-Cath Suture Anchor Delivery Catheter — Evaluate changes in emptying, hormones, satiety and weight loss with use of the g-Cath Suture Anchor Delivery Catheter in maximizing g-Cath Suture Anchor placement to as high as 25 anchors.

SUMMARY:
The purpose of this study is to help find out more about how the Primary Obesity Surgery Endoluminal (POSE) procedure makes patients feel less hungry and fuller faster, leading to weight loss. In this study, USGI Medical wants to see if stomach emptying and gastro-intestinal hormone levels change after a POSE procedure with an increased (as compared to typical) number of anchors placed.

DETAILED DESCRIPTION:
This study will use the USGI Medical Incisionless Operating Platform (IOP) to determine the affects of placing more Suture Anchors per patient (as compared to the current practice) in Primary Obesity Surgery Endoluminal(POSE). USGI wants to see if placing more anchors (particularly in the distal body/antrum region) significantly impacts primary weight loss, satiety, and metabolic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Has a BMI of >30 and <40
* Male or female ≥21 yrs. of age and < 60 yrs. of age at time of enrollment
* Patient has had no significant weight change (+/- 5% of total body weight) in last 6 months but has been able to lose significant weight in the past with diet and exercise.
* Is a reasonable candidate for general anesthesia
* Agrees not to have any additional weight loss interventional procedures or liposuction for at least 18 months following study enrollment and agrees not to take any prescription or over the counter weight loss medications for at least 1 year.
* Physically and mentally able to comply with the visit schedule, ancillary testing, and behavior modification (diet and exercise) required for the study and agrees to study commitment requirements
* Had successful completion of the pre-screening, nutritional and educational programs and psychological assessment supporting that the subject is an appropriate bariatric surgical candidate

Exclusion Criteria:

* History of (or intra-operative evidence of) bariatric, gastric or esophageal surgery
* Esophageal stricture or other anatomy and/or condition that could preclude passage of endolumenal instruments
* Moderate to severe Gastro-esophageal reflux disease (GERD)
* Known hiatal hernia >3cm by history or as determined by UGI exam or endoscopy
* Known GI motility disorder or pancreatic insufficiency/disease
* Intra-operative Exclusion: Active peptic ulcer or hiatal hernia >3cm
* Pregnancy.
* Present Corticosteroid Use
* History of inflammatory disease of GI tract
* Severe coagulopathies, hepatic insufficiency or cirrhosis
* History or present use of insulin or insulin derivatives for treatment of diabetes
* Had Type II Diabetes Mellitus (as defined by HgbA1c >6.0) for greater than 2 years at the time of enrollment
* Uncontrolled Type II DM (HgbA1c >7.0 at screening)
* Patient has quit smoking within last 6 months at time of enrollment or plans to quit smoking in the next year
* Patient has a history of drug or alcohol abuse or actively abusing either
* Patient is presently being treated with medication for depression, psychosis, or other mood or eating disorder
* Non-ambulatory or has significant impairment of mobility
* Works for, or is first degree relative of investigator, study institution, or support staff involved in the study.
* Known hormonal or genetic cause for obesity
* Participating in another clinical study
* Patient is on medications known to impact GI motility or gut hormones that cannot be discontinued prior to nuclear testing
* Have work hours, family obligations or transportation issues that could interfere with patient returning for all scheduled evaluations, tests and nutritional counseling.
* Lives >60 kilometers from investigator site.
* Patient is not able to provide written informed consent

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 18 months
  Weight loss will be monitored and recorded on a monthly basis for up to 18 months post POSE with the proportion of subjects achieving ≥25% excess weight loss (EWL) at 12 months (Met Life criteria)being the primary efficacy endpoint

SECONDARY OUTCOMES:
Gastric emptying | Immediately Pre-procedure, & 2 & 6 months post procedure
  This test consists of determining if there is a Clinically significant change in the duration of a radioactive marker (which is non-absorbable, and free of any food components) in a stomach pre and post POSE. In order to carry out this test, a piece of food is marked with a radioactive isotope and, by using an abdominal gamma camera; detections of radioactivity are made in the stomach during the postprandial period.

OTHER OUTCOMES:
Satiety | Immediately Pre-procedure, & 2 & 6 months post procedure
  This test consists of determining if there is a Clinically significant change in Satiety pre and post POSE. The subjects ingest a nutritional drink (Ensure) at a constant rate of 30 mL per minute, constantly filling the glass with a perfusion pump (Gemini PC-2, IMED, San Diego, CA). (The subjects are not conscious of the volume being ingested.) The subjects are instructed to maintain consumption at the fill rate. Participants take note of their sensation of satiety with a graphical classification scale, which combines verbal descriptors on a scale of 0 to 5 (0 = no symptoms, 1 = first sensation of fullness [threshold]; 2 = light, 3 = moderate, 4 = severe, and 5 = maximum fullness or unbearable). The participants are told to stop taking the food product when a score of 5 is obtained. The maximum consumption of volume of the nutritional drink is recorded.
Peptide Measurements | Immediately Pre-procedure & 2 Months post procedure
  This test consists of determining if there is a Clinically significant change in peptides pre and post procedure.
  1. Samples to be collected when fasting and 30, 60, 90, and 120 minutes after a standard meal (A meal consisting of 400 calories is used), The meal must be consumed within 10 minutes.
  2. Samples to be collected by ELISA are: C-peptide, serum insulin, glucose, PYY, GLP-1 (active), leptin, and GIP. Total ghrelin level to be analyzed by RIA.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge C Espinos, MD, Principal Investigator — Centro Medico Teknon
Locations (1):
- Centro Medico Teknon, Barcelona, Spain